CLINICAL TRIAL: NCT00285415
Title: A Phase II Evaluation of Docetaxel and Carboplatin Followed by Tumor Volume Directed Pelvic Plus or Minus Para-Aortic Irradiation for Stage III/IV Endometrial Carcinoma
Brief Title: A Phase II Evaluation of Docetaxel and Carboplatin Followed by Tumor Volume Directed Pelvic Irradiation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator abruptly left Carilion.
Sponsor: Carilion Clinic (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EndoRT; WIRB PRO NUM: 20050247 (Other: Western Institutional Review Board)
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Advanced Endometrial Adenocarcinoma, Stage III A, B, C
Keywords: Advanced endometrial adenocarcinoma, stage III A, B, C
MeSH Terms: interventions — Docetaxel; Carboplatin

ARMS (1):
- Doc and Car (Other): Receiving Doc and Car
  Interventions: Drug: Docetaxel and Carboplatin

INTERVENTIONS:
Drug: Docetaxel and Carboplatin — docetaxel (75 mg/m2) + carboplatin (AUC 6) IV every 3 weeks X 6 cycles

SUMMARY:
The purpose of this study is to determine the effectiveness of the combination of the two drugs, docetaxel (Taxotere®) and carboplatin (Paraplatin®) followed by radiation directed at the tumor in treating your endometrial cancer.

DETAILED DESCRIPTION:
Endometrial carcinoma is the most common malignancy in the female reproductive tract. For the percentage of patients with advanced stage (III - IV) optimum adjuvant therapy status-post surgical staging and/or optimal cytoreductive surgery is not well defined and limited in the rates of response. Survival rates range from 18 - 49% with high levels of toxicity with the current treatment regimens.

The Gynecologic Oncology Group (GOG) explored the use of chemotherapy in protocol #107 comparing adriamycin with a combination of adriamycin and cisplatin. This trial boasted a 45% response rate for the combination arm compared to a 27% response rate in the adriamycin only arm. Although no difference was seen in overall survival, the combination arm showed an improvement in progression free survival from 3.8 to 5.7 months. Subsequently, GOG protocol #122 randomized patients to this chemotherapeutic regimen versus whole abdominal radiation therapy. This trial is now closed to accrual and results are pending.

Ball et. al. reported on a phase II trial of paclitaxel in advanced or recurrent endometrial cancer done through the GOG.(3) At 250 mg/m2 (200mg/m2 for patients with previous radiation therapy) over 24 hours, every 21 days, 10/28 patients responded. There were 4 complete responders and 6 partial responders with an overall response rate of 35.7%. Toxicity was remarkably high with grade 3 and 4 neutropenia and neurotoxicity seen in 62% and 10.7%, respectively.

Dimpoulos et. al. reported the use of paclitaxel 175 mg/m2 over 3 hours and cisplatin 75mg/m2 every 21 days in advanced or recurrent endometrial carcinoma.(4) A 67% objective response rate was seen with 29% showing a complete response and 38% partial response. Toxicities included a 9% grade 3 and 4 peripheral neuropathy rate. These response rates changed the standard of care in the community setting from the more toxic regimen of adriamycin and cisplatin to paclitaxel and carboplatin.

Hoskins et. al. substituted carboplatin for cisplatin in an effort to reduce the peripheral neuropathy seen in the Dimpoulos trial. This phase II combination of paclitaxel and carboplatin with radiation therapy in advanced endometrial cancer resulted in a 75% response rate. The median failure-free survival time was 23 months, with a 62% 3-year overall survival rate. Toxicities were primarily hematologic and reversible.

The ongoing GOG protocol, #184, is exploring the combination of tumor directed radiation followed by a randomization to adriamycin and cisplatin versus adriamycin, cisplatin and paclitaxel with G-CSF support. Increased toxicity will be expected in the three-drug regimen. With a significant response rates to a combination of paclitaxel and carboplatin along with radiation therapy in the phase II setting it is hard to justify the added toxicity of this three-drug regimen.

The SCOTROC phase III trial comparing docetaxel (75 mg/m2) over 1 hour plus carboplatin (AUC 6) vs. paclitaxel (175 mg/m2) over 3 hours plus carboplatin (AUC 6) yielded equivalent overall response rates in 1,077 patients with ovarian cancer. The docetaxel arm resulted in significantly less overall grade 2 and 3 sensory and motor neurotoxicity. Only 4 patients withdrew from the trial due to neurotoxicity on the docetaxel arm vs. 32 patients on the paclitaxel arm. However, the docetaxel arm resulted in a higher incidence of neutropenia and associated complications without compromising treatment delivery of overall safety.

Based on the information to date, it seems prudent to explore a phase II trial of docetaxel plus carboplatin every 3 weeks for 6 cycles followed by radiation therapy in the management of patients with advanced endometrial cancer. The proposed protocol design requires that chemotherapy be administered prior to radiation therapy in order to control distant metastatic disease before attempting to control for local-regional recurrences with radiation.

ELIGIBILITY:
Inclusion Criteria:

* All patients with advanced endometrial adenocarcinoma, stage III A, B, C and Stage IV confined to the pelvis, and recurrent disease limited to the pelvis.
* Surgical stage III and limited stage IV disease, including those patients with positive adnexa, tumor invading the serosa, positive and/or para-aortic nodes, pelvic metastases, positive pelvic washings or vaginal involvement.
* Histology must be adenocarcinoma, adenosquamous cell, squamous cell, clear cell or serous papillary carcinoma
* Status post surgical resection, including a hysterectomy and bilateral salpingo-oophorectomy within the past
* 6 weeks (Pelvic lymph node and para-aortic lymph node sampling are optional)
* Patients may be sub-optimally or optimally debulked (disease < 2 cm). Patients are eligible with measurable disease or evaluable
* disease. All positive para-aortic node patients must be further staged by chest CT scan. If chest CT scan is negative, patients are eligible.
* Patients who have met the pre-entry criteria including following lab findings:

  * ANC > 1500, Platelet count > 100,000/mm3, Hemoglobin ≥ 8 mg/dl, Creatinine < 2.0 mg/dl.
  * Total Bilirubin must be within normal limits. (WNL)
  * AST or ALT and Alkaline Phosphatase must be within the range allowing for eligibility
  * Patients who have signed an approved informed consent.
  * GOG Performance Grade 0, 1, or 2.
  * Women ≥ 18 years of age

Exclusion Criteria:

* Patients with Stage IV or recurrent disease outside of the pelvis.
* Patients who have had prior pelvic or abdominal radiation therapy.
* Patients with concomitant malignancy other than non-melanoma skin cancer.
* Patient with a prior malignancy who have been disease-free for < 5 years or who received prior chemotherapy or radiation therapy for that malignancy.
* Patients with a history of serious co-morbid illness that would preclude protocol therapy.
* Patients with an estimated survival of less than three months.
* Patients with parenchymal liver metastases.
* Patients who received prior chemotherapy excluding low-dose methotrexate for rheumatologic reasons.
* Histology consistent with uterine sarcomas, carcinosarcoma or leiomyosarcoma.
* Women with baseline peripheral neuropathy Grade ≥ 2.
* Women with a history of severe hypersensitivity reaction to drugs formulated with polysorbate 80.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2005-04 (Actual); Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) for patients treated with docetaxel and carboplatin as measured by RECIST 1.1 | every 3 months
  to estimate the overall response rate (ORR) for women with newly diagnosed stages III-IV or recurrent endometrial carcinoma treated with docetaxel and carboplatin followed by tumor volume directed pelvic plus or minus para-aortic irradiation.

SECONDARY OUTCOMES:
Progressive free survival (PFS) for patients treated with docetaxel and carboplatin as measured by CA125. | every 3 months for 2 years and then every 6 months for 3 years. Yearly after 5 years.
  To estimate the progressive free survival (PFS)
To estimate overall survival (OS) | every 3 months for 2 years then every 6 months for 3 years
  To estimate overall survival (OS)
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 5 years
  Determine the safety and tolerability of docetaxel and carboplatin

CONTACTS AND LOCATIONS:
Overall Officials: Dennis R Scribner, JR, MD, Principal Investigator
Locations (2):
- United States (2):
  - Gynecologic Oncology Research & Development, LLC, Greenville, South Carolina
  - Carilion GYN Oncology Associates, Roanoke, Virginia